CLINICAL TRIAL: NCT05176665
Title: Phase Ib/II, Open-Label Study of EMB-01 in Patients With Advanced/Metastatic Gastrointestinal Cancers
Brief Title: EMB-01 in Patients With Advanced/Metastatic Gastrointestinal Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai EpimAb Biotherapeutics Co., Ltd. (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB01X201
Record Dates: First submitted 2021-11-03; First posted 2022-01-04 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms; Neoplasm Metastasis; Metastatic Gastrointestinal Carcinoid Tumor
Keywords: Human Bispecific antibody; Epidermal Growth Factor Receptor (EGFR); c-Mesenchymal-Epithelial Transition (cMet); Neoplasms， Neoplasm Metastasis; Neoplasm Metastasis; EMB-01，Tyrosine Kinase Inhibitor (TKI) Resistant
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase Ib and Phase II (Experimental): The study will consist of Phase Ib and Phase II. The study is planning to recruit approximately 152 patients in total for advanced/metastatic GI cancers, which include 24 patients in Phase Ib and up to approximately 128 patients in Phase II. For GC, HCC, and BTC groups, up to approximately 24 patients may be enrolled in Phase Ib and Phase II. For CRC group, up to approximately 80 patients may be enrolled in Phase Ib and Phase II with up to 40 patients in each subgroup.
  Interventions: Drug: EMB-01

INTERVENTIONS:
Drug: EMB-01 — EMB-01 at the RP2D of 1600 mg will be administered as an IV infusion once weekly (QW) throughout the study. One cycle is defined as 4 weeks (4 doses).
  Other Names: FIT-013a

SUMMARY:
This study is to evaluate the safety and antitumor activity of EMB-01 in advanced/metastatic gastrointestinal cancers, including gastric cancer, hepatocellular cancer, cholangiocarcinoma and colorectal cancer.

DETAILED DESCRIPTION:
This is an open-label, Phase Ib/II, multi-stage study of EMB-01 in patients with advanced gastrointestinal tumors including gastric cancer, hepatocellular cancer, cholangiocarcinoma cancer and colorectal cancer, who have EGFR/cMET gene alterations or protein over expression and progressed on available standard therapies and for whom no standard therapy exists that would confer clinical benefit. All patients will be prescreened for cMET and EGFR genetic alterations and protein expression. Only those who met the molecular pre-screening criteria will proceed to clinical screening to determine the eligibility. The study will consist of Phase Ib part and Phase II part, both phases will consist of a molecular prescreening period, screening period, treatment period, safety follow-up period, and disease progression follow-up.

ELIGIBILITY:
Inclusion Criteria:

Molecular Pre-screening Inclusion criteria

1. cMET amplification in tumor sample; OR
2. cMET overexpression in tumor sample; OR
3. EGFR overexpression in tumor sample; OR
4. Other EGFR or cMET gene alteration in blood sample (circulating tumor DNA, ctDNA).

In Phase II, CRC patients must provide blood sample for NGS test, but may not provide tumor samples at prescreening visit. CRC patients don't need to meet the above criteria of EGFR/cMET amplification, overexpression or gene aberration.

Screening Inclusion Criteria

1. Able to understand and willing to sign the Informed Consent Form (ICF).
2. Histologically/cytologically confirmed advanced/metastatic gastric cancer, HCC, BTC, and colorectal cancer with measurable disease (RECIST V1.1). To be eligible, patients must meet following criteria:

   1. Have failed all standard of care therapies known to confer clinical benefit. Patients who is not tolerable on standard of care therapies, or no standard of care therapies available, or refused standard of care therapies are eligible.
   2. Have measurable disease as defined by RESIST v 1.1.
3. Archival tumor tissue (formalin-fixed or paraffin-embedded, collected within 1 year) or a new biopsy collected in the molecular pre-screening visit.
4. Must have adequate organ function.
5. Regarding prior anti-tumor therapy:

   1. Patients who have received any anticancer drugs approved or investigational, including chemotherapy, immune therapy, hormonal therapy (Exceptions: hormone-replacement therapy, testosterone or oral contraceptives), biologic therapy, must have stopped treatment at least 4 weeks or within 5 half -lives whichever shorter before first dose of EMB-01.
   2. Local radiotherapy or radiation therapy for bone metastases must have stopped 2 weeks before first dose of EMB-01. No therapeutic radiopharmaceuticals are taken within 8 weeks before first dose of EMB-01.
   3. Patients who have received prior targeted therapies must have stopped treatment for at least 4 weeks or within 5 half-lives, whichever is shorter before first dose of EMB-01.
6. Female patient with fertility or male patient whose partner has fertility should use one or more contraceptive methods for contraception starting from screening period and continue throughout the study treatment and for 3 months.
7. ECOG score ≤1.

Exclusion Criteria:

Molecular Pre-screening Exclusion Criteria

Subject who meets any of the following criteria can't be proceeded to clinical screening:

1. Patients who are unwilling to sign the molecular pre-screening ICF.
2. Patients for whom the results of central laboratory testing do not meet the molecular pre-screening inclusion criteria.
3. Patients with a documented gene alteration including but not limited to HER2, KRAS, NRAS, BRAF, NTRK, ALK, RET, ROS1, and FGFR, etc. that is known to confer resistance to EGFR and/or cMET inhibitors.* * In Phase II, CRC patients with activated KRAS, NRAS or BRAF mutation should be excluded, but patients with other gene alterations do not need to be excluded.

Screening Exclusion Criteria

1. Life expectancy < 3 months.
2. Patients with primary central nervous system (CNS) malignancy or symptomatic CNS (leptomeningeal or brain) metastases are not allowed. Patients with asymptomatic CNS metastases are eligible.
3. Pregnant or nursing females.
4. Patients who have had major surgery within the 28 days from the screening. Surgical wounds must be completely healed.
5. Any other serious underlying medical (e.g. uncontrolled diabetes mellitus, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, cardiac conditions), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0 | Phase 1b, screening up to follow-up (30 days after the last dose)
  Number of participants with Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0
Best Overall Response (BOR) as assessed by RECIST v1.1 | Phase II, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Best Overall Response (BOR) as assessed by RECIST v1.1
Objective Response Rate (ORR) as assessed by RECIST v1.1 | Phase II, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Objective Response Rate (ORR) as assessed by RECIST v1.1
Duration of Response (DoR) as assess by RECIST v1.1 as assess by RECIST v1.1 | Phase II, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Duration of Response (DoR) as assess by RECIST v1.1 as assess by RECIST v1.1
Disease Control Rate (DCR) as assess by RECIST v1.1 | Phase II, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Disease Control Rate (DCR) as assess by RECIST v1.1
Progression-Free Survival (PFS) as assess by RECIST v1.1 | Phase II, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Progression-Free Survival (PFS) as assess by RECIST v1.1
Maximum serum concentration (Cmax) of EMB-01 | Phase Ib only, up to 3 months after first study drug administration
  Maximum serum concentration (Cmax) of EMB-01
Trough serum concentration (Ctrough) of EMB-01 | Phase Ib only, predose, through treatment completion, an average of 1 year
  Trough serum concentration (Ctrough) of EMB-01
Area under the concentration-time curve from time 0 (pre-dose) to the time of the dosing interval (AUC0-t) | Phase Ib only, up to 3 months after first study drug administration
  Area under the concentration-time curve from time 0 (pre-dose) to the time of the dosing interval (AUC0-t)
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | Phase Ib only, up to 3 months after first study drug administration
  Area under the concentration-time curve from time 0 to infinity (AUC0-inf)
Elimination half-life (T1/2) | Phase Ib only, up to 3 months after first study drug administration
  Elimination half-life (T1/2)
Systemic clearance (CL) | Phase Ib only, up to 3 months after first study drug administration
  Systemic clearance (CL)
Apparent volume of distribution at steady-state (Vss) | Phase Ib only, up to 3 months after first study drug administration
  Apparent volume of distribution at steady-state (Vss)
Accumulation Ratio (AR) after multiple dosing | Phase Ib only, up to 3 months after first study drug administration
  Accumulation Ratio (AR) after multiple dosing
Incidence of positive ADA | Phase Ib only, up to the 30-day safety follow-up visit after EOT
  Incidence of positive ADA
Clinical benefit rate(CBR) as assess by RECIST v1.1 | Phase II, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Clinical benefit rate(CBR) as assess by RECIST v1.1

SECONDARY OUTCOMES:
Number of participants with Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0 | Phase II, screening up to follow-up (30 days after the last dose)
  Number of participants with Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0
Maximum serum concentration (Cmax) of EMB-01 | Phase II, up to 3 months after first study drug administration
  Maximum serum concentration (Cmax) of EMB-01
Trough serum concentration (Ctrough) of EMB-01 | Phase II, predose, through treatment completion, an average of 1 year
  Trough serum concentration (Ctrough) of EMB-01
Incidence of positive ADA | Phase II , up to the 30-day safety follow-up visit after EOT
  Incidence of positive ADA
Best Overall Response (BOR) as assessed by RECIST v1.1 | Phase Ib, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Best Overall Response (BOR) as assessed by RECIST v1.1
Objective Response Rate (ORR) as assessed by RECIST v1.1 | Phase Ib, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Objective Response Rate (ORR) as assessed by RECIST v1.1
Duration of Response (DoR) as assess by RECIST v1.1 as assess by RECIST v1.1 | Phase Ib, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Duration of Response (DoR) as assess by RECIST v1.1 as assess by RECIST v1.1
Disease Control Rate (DCR) as assess by RECIST v1.1 | Phase Ib, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Disease Control Rate (DCR) as assess by RECIST v1.1
Progression-Free Survival (PFS) as assess by RECIST v1.1 | Phase Ib, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Progression-Free Survival (PFS) as assess by RECIST v1.1
Clinical benefit rate(CBR) as assess by RECIST v1.1 | Phase Ib, from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Clinical benefit rate(CBR) as assess by RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (14):
- MD Anderson Cancer Center, Houston, Texas, United States
- China (13):
  - Beijing cancer Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Gansu Provincial Hospital, Lanzhou
  - The Affiliated hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No